CLINICAL TRIAL: NCT05274321
Title: Efficacy of the Nanodropper Device on Pupillary Dilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Nanodropper, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-32530-OBS
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Results first posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Dilation
MeSH Terms: conditions — Dilatation, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Pediatric Participant's Eyes Using Standard Pupilary Dilation (Active Comparator): Consenting pediatric participants will undergo standard pupillary dilation in one eye.
  Interventions: Device: Standard Eye Dropper
- Pediatric Participant's Eyes using Nanodropper attachment (Experimental): Consenting pediatric participants will undergo pupillary dilation in the second eye using the Nanodropper attachment.
  Interventions: Device: Nanodropper

INTERVENTIONS:
Device: Nanodropper — Device used for administering eye drops
  Arms: Pediatric Participant's Eyes using Nanodropper attachment
Device: Standard Eye Dropper — Standard Eye Dropper used for administering eye drops
  Arms: Pediatric Participant's Eyes Using Standard Pupilary Dilation

SUMMARY:
Prescription eye drop bottles elute drops that exceed the capacity of the human eye by five times. This study describes performing in clinic dilation using a novel solution for combating medical waste with Nanodropper, an eye drop bottle adapter that creates smaller eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Participants under the age of 18 years old

Exclusion Criteria:

* Participants 18 years and older
* Pupillary or anterior segment abnormality
* Participants with pre-existing health conditions that would prevent pupillary dilation.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Oatts, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children 18 years of age or younger undergoing pupillary dilation as part of a routine eye examination at the University of California, San Francisco, at the Pediatric Ophthalmology Clinic between August 4, 2021, and November 19, 2021 were assessed for eligibility. Children who did not show up to appointments or did not meet inclusion criteria were not enrolled in the study.
Units Other Than Participants: eyes
Groups:
- Eyes Recieving Eye Drops From Standard of Care: Each participant was randomized to receive eye drops using the standard of care dropper in one of their eyes
- Eyes Recieving Eye Drops Using Nanodropper Device: Each participant was randomized to receive eye drops using the Nanodropper adaptor in one of their eyes.
  The Nanodropper device is an eye drop adaptor that administers a smaller quantity (10.4 ml) of eye drops
Period: Overall Study
Arm/Group | Eyes Recieving Eye Drops From Standard of Care | Eyes Recieving Eye Drops Using Nanodropper Device
Started | 50; 50 eyes | 50; 50 eyes
Completed | 50; 50 eyes | 50; 50 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were determined for participants who enrolled in the study and cooperated with all measurements.
Groups:
- Pediatric Participants: Consenting participants will undergo standard pupillary dilation in one eye and pupillary dilation in the second eye using the Nanodropper attachment.
  Nanodropper: Device used for administering eye drops
Arm/Group | Pediatric Participants
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Spherical Equivalent
Description: Cycloplegia is the paralysis of the ciliary muscle of the eye resulting in dilatation of the pupil and paralysis of accommodation.
  Cycloplegia is defined as the "change score." Change scores were calculated by subtracting the spherical equivalent value after dilation from the value before dilation for each eye.
Time Frame: Before dilation and 30 minutes after dilation
Population: Participants received eye drops from the Nanodropper in one eye only and Standard of Care in the other eye.
Measure: Mean (95% Confidence Interval); unit: Diopters
Units Other Than Participants: Eye
Arm/Group | Eyes Recieving Eye Drops From Standard of Care | Eyes Recieving Eye Drops Using Nanodropper Device
Number analyzed (Participants) | 50 | 50
Number analyzed (Eye) | 50 | 50
Diopters
  Before Dilation | -2.62 [-3.59 to -1.65] | -2.28 [-3.17 to -1.39]
  After Dilation | -0.86 [-1.75 to 0.03] | -0.55 [-1.43 to 0.34]
  Change Score | 1.76 [1.11 to 2.41] | 1.73 [1.11 to 2.36]
Statistical Analysis 1: Comparison: Eyes Recieving Eye Drops From Standard of Care vs Eyes Recieving Eye Drops Using Nanodropper Device; Absolute between-eye differences were calculated for each participant by subtracting the standard of care (SOC) change score from the Nanodropper change score. The confidence interval (CI) is 95%; Test type: Non-Inferiority — The noninferiority margin was determined by taking 10% of the standard of care change score. Noninferiority was determined for each outcome if the noninferiority margin did not overlap with the regression coefficient's 95% confidence interval; p = 0.22, Regression, Linear — Wald P values were calculated by testing whether the regression coefficient met or exceeded the noninferiority margin; The threshold for significance is 0.0167

2. Primary Outcome: Maximum Pupil Diameter
Description: The pupil is the opening in the center of the iris (the structure that gives our eyes their color). The diameter is a straight line passing from side to side through the center of the pupil, which is shaped like a circle.
Time Frame: Before dilation and 30 minutes after dilation
Population: Participants received eye drops from the Nanodropper in one eye only and Standard of Care in the other eye.
Measure: Mean (95% Confidence Interval); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Eyes Recieving Eye Drops From Standard of Care | Eyes Recieving Eye Drops Using Nanodropper Device
Number analyzed (Participants) | 50 | 50
Number analyzed (Eyes) | 50 | 50
mm
  Before Dilation | 5.95 [5.76 to 6.14] | 6.01 [5.80 to 6.22]
  After Dilation | 7.91 [7.72 to 8.10] | 7.81 [7.61 to 8.01]
  Change Score | 1.95 [1.77 to 2.13] | 1.77 [1.58 to 1.96]
Statistical Analysis 1: Comparison: Eyes Recieving Eye Drops From Standard of Care vs Eyes Recieving Eye Drops Using Nanodropper Device; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The noninferiority margin was determined by taking 10% of the standard of care change score. Noninferiority was determined for each outcome if the noninferiority margin did not overlap with the regression coefficient's 95% confidence interval; p = 0.02, Regression, Linear — Wald P values were calculated by testing whether the regression coefficient met or exceeded the noninferiority margin; The threshold for significance is 0.0167

3. Primary Outcome: Constriction Percentage
Description: Pupillary constriction percentage was calculated by the pupillometer in response to a 180-micro watt flash: (maximum - minimum) / maximum
Time Frame: Before and 30 minutes after dilation
Population: Participants received eye drops from the Nanodropper in one eye only and Standard of Care in the other eye.
Measure: Mean (95% Confidence Interval); unit: percent change
Units Other Than Participants: Eyes
Arm/Group | Eyes Recieving Eye Drops From Standard of Care | Eyes Recieving Eye Drops Using Nanodropper Device
Number analyzed (Participants) | 50 | 50
Number analyzed (Eyes) | 50 | 50
percent change
  Before Dilation | 30.44 [28.95 to 31.93] | 31.07 [29.53 to 32.61]
  After Dilation | 5.67 [3.21 to 8.14] | 6.26 [4.35 to 8.17]
  Change Score | -24.76 [-27.53 to -22.00] | -24.81 [-26.72 to -22.49]
Statistical Analysis 1: Comparison: Eyes Recieving Eye Drops From Standard of Care vs Eyes Recieving Eye Drops Using Nanodropper Device; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.03, Regression, Linear — Wald P values were calculated by testing whether the regression coefficient met or exceeded the noninferiority margin; The threshold for significance is 0.0167

4. Secondary Outcome: Change in Intraocular Pressure
Description: Intraocular pressure is the pressure, or force, inside of your eyes. Specifically, it's a measurement of the fluid pressure in your aqueous humor.
Time Frame: Before and 30 minutes After Dilation
Measure: Mean (95% Confidence Interval); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Eyes Recieving Eye Drops From Standard of Care | Eyes Recieving Eye Drops Using Nanodropper Device
Number analyzed (Participants) | 50 | 50
Number analyzed (eyes) | 50 | 50
mmHg
  Before Dilation | 17.36 [16.24 to 18.48] | 18.13 [17.11 to 19.16]
  After Dilation | 18.42 [17.31 to 19.53] | 17.96 [16.84 to 19.08]
  Change Score | 1.06 [-0.08 to 2.20] | -0.17 [-1.28 to 0.93]
Statistical Analysis 1: Comparison: Eyes Recieving Eye Drops From Standard of Care vs Eyes Recieving Eye Drops Using Nanodropper Device; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.25, Regression, Linear — Wald P values were calculated by testing whether the regression coefficient met or exceeded the noninferiority margin; The threshold for significance is 0.0167

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the time of the participant visit. Each participant visit lasted on average 1 hour.
Description: Study staff monitored participants for adverse effects including transient seizure, psychosis, subjective fever, and subjective tachycardia.
Arm/Group | Eyes Recieving Eye Drops From Standard of Care | Eyes Recieving Eye Drops Using Nanodropper Device
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
We chose a noninferiority margin of a loss of 10% of the treatment effect, which is more conservative than the 50% margin that has been recommended for some industry trials by the United States Food and Drug Administration. Study staff and participants were not masked to the intervention. Additionally, this cohort comprised predominantly children with dark irides but could limit the generalizability of these results. We did not measure minimizing systemic side effects and local irritation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT05274321/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT05274321/ICF_001.pdf